CLINICAL TRIAL: NCT00133939
Title: Proportional Ventilation and Ventilatory Synchronism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2004.359
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Mechanical Ventilation
Keywords: Proportional assisted ventilation; Pressure support ventilation; Synchronism during mechanical ventilation; Patients undergoing partial mechanical ventilation
MeSH Terms: interventions — Respiration, Artificial

INTERVENTIONS:
Procedure: Mechanical ventilation

SUMMARY:
Synchronism of gas flow delivered by the ventilator and muscular effort of the patient will be studied during two kinds of ventilation. The first one is the proportional assisted ventilation during which the gas flow is theoretically adapted to the patient's muscular effort within the breath. The second is the pressure support ventilation during which the gas flow is delivered to maintain the inspiratory pressure stable. The hypothesis is that the first mode allows a better synchronism.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing partial ventilatory support

Exclusion Criteria:

* Patients failing the weaning process

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10

PRIMARY OUTCOMES:
Time lag between the onset of diaphragmatic electromyogram (EMG) signal and the zero crossing of the inspiratory flow, over five minutes

SECONDARY OUTCOMES:
Number per minute of failing breaths: breath with muscular effort without any inspiratory flow

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul VIALE, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Background] Ganne O, Abisseror M, Menault P, Malhiere S, Chambost V, Charpiat B, Ganne C, Viale JP. Low-dose ketamine failed to spare morphine after a remifentanil-based anaesthesia for ear, nose and throat surgery. Eur J Anaesthesiol. 2005 Jun;22(6):426-30. doi: 10.1017/s0265021505000724. PMID 15991504
- [Background] Mechet I, Lhuillier F, Blanchet MC, Pouyet M, Viale JP, Goudable J, Annat G, Scoazec JY, Boillot O, Liotard D, Merle E, Delafosse B. Liver function during extracorporeal whole liver perfusion in a pig model of acute ischemic liver failure. ASAIO J. 2004 Sep-Oct;50(5):503-11. doi: 10.1097/01.mat.0000136509.08283.b9. PMID 15497393